CLINICAL TRIAL: NCT03476356
Title: L-Carnitine and Clomiphene Citrate for Induction of Ovulation in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Rehab Mohamed Abdelrahman, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCO L
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene

STUDY DESIGN:
Intervention Model Description: A total of 106 women with the diagnosis of PCOS based on the European Society of Human Reproduction and Embryology/ American Society for Reproductive Medicine (ESHRE/ASRM) guidelines criteria (Rotterdam Criteria, 2003) will be randomly assigned using a computer-generated randomization sheet and they will be distributed into two groups:
  Group L (53 patients):
  This group will receive oral clomiphene citrate (Clomid, Global Napi Pharmaceuticals (GNP), Egypt) (50 mg tablet, two times per day) from the third day of the cycle until the seventh day of the cycle plus oral carnitine supplementation (Carnivita Forte, Eva Pharma, Egypt) (1g tablet, three times per day) from the third day of the cycle until the day of the pregnancy test.
  Group C (53 patients):
  This group will receive oral clomiphene citrate only (Clomid, Global Napi Pharmaceuticals (GNP), Egypt) (50 mg tablet, two times per day) from the third day of the cycle until the seventh day of the cycle.
Who Masked: Participant, Care Provider
Masking Description: One hundred and six opaque envelopes will be numbered serially and, in each envelope, there will be the corresponding letter which denotes the allocated group according to the randomization table. Then all of the envelopes will be closed and they will be placed in one box. When the first woman arrives, the first envelope will be opened and she will be allocated according to the letter inside, and this step will be repeated until the 106 envelopes are finished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Experimental): This group will receive oral clomiphene citrate (Clomid, Global Napi Pharmaceuticals (GNP), Egypt) (50 mg tablet, two times per day) from the third day of the cycle until the seventh day of the cycle plus oral carnitine supplementation (Carnivita Forte, Eva Pharma, Egypt) (1g tablet, three times per day) from the third day of the cycle until the day of the pregnancy test.
  Interventions: Drug: oral clomiphene citrate; Drug: oral carnitine supplementation
- Group C (Active Comparator): This group will receive oral clomiphene citrate only (Clomid, Global Napi Pharmaceuticals (GNP), Egypt) (50 mg tablet, two times per day) from the third day of the cycle until the seventh day of the cycle.
  Interventions: Drug: oral clomiphene citrate

INTERVENTIONS:
Drug: oral clomiphene citrate — oral clomiphene citrate 50 mg tablet, two times per day will be received from the third day of the cycle until the seventh day of the cycle.
  Other Names: clomid
Drug: oral carnitine supplementation — oral carnitine supplementation 1g tablet, three times per day will be received from the third day of the cycle until the day of the pregnancy test.
  Other Names: Carnitiva Forte
  Arms: Group L

SUMMARY:
The purpose of the study to assess the efficacy of adding L-carnitine to clomiphene citrate for increasing the ovulation and the pregnancy rate in women with PCOS.

DETAILED DESCRIPTION:
A total of 106 women with the diagnosis of PCOS based on the European Society of Human Reproduction and Embryology/ American Society for Reproductive Medicine (ESHRE/ASRM) guidelines criteria (Rotterdam Criteria, 2003) will be randomly assigned using a computer-generated randomization sheet and they will be distributed into two groups:

1. Group L (53 patients):

   This group will receive oral clomiphene citrate (Clomid, Global Napi Pharmaceuticals (GNP), Egypt) (50 mg tablet, two times per day) from the third day of the cycle until the seventh day of the cycle plus oral carnitine supplementation (Carnivita Forte, Eva Pharma, Egypt) (1g tablet, three times per day) from the third day of the cycle until the day of the pregnancy test.
2. Group C (53 patients):

This group will receive oral clomiphene citrate only (Clomid, Global Napi Pharmaceuticals (GNP), Egypt) (50 mg tablet, two times per day) from the third day of the cycle until the seventh day of the cycle. Serum FSH, LH & free testosterone concentrations will be measured on day 3 (basal) of the cycle. Trans-vaginal folliculometry will be performed on all women on days 7 and 9 of the cycle and then individualized according to the response. When one leading follicle attains a diameter of 17mm or more, the endometrial thickness will be measured and 10,000 IU of Human chorionic gonadotropin (hCG) will be given (im injection; Pregnyl, organon, Holland). Timed intercourse will be advised after 36-48 hours from the night of hCG administration for 2 successive days. Ovulation success will be confirmed by transvaginal ultrasound which will show that the leading follicle has collapsed, and some fluid appeared in the Douglas pouch.

Serum progesterone will be measured on day 8 post hCG injection, ovulation will be confirmed if the serum progesterone level is ≥ 5 ng/ml (Leiva et al., 2015).

Luteal-phase support will not be provided in both groups. Pregnancy test will be done in the form of testing the level of beta hCG in the blood after 14 days once the success of the ovulation process has been confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18-35 years.
2. Normal Hysterosalpingo-graphy (HSG).
3. Normal Semen analysis of the husband.
4. Diagnosed with PCOS based on the (ESHRE/ASRM) guidelines criteria (Rotterdam Criteria 2003).

Exclusion Criteria:

1. Patient's refusal.
2. Male factors of infertility and/or abnormal HSG.
3. Hyperprolactinemia (prolactin ≥ 22 ng/dl).
4. FSH on day 3 > 15 mIU/mL.
5. Gross ovarian pathology diagnosed by ultrasound.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Ovulation success by trans-vaginal ultrasound | 36-48 hours after night of hCG administration
  Ovulation success will be confirmed by transvaginal ultrasound which will show that the leading follicle has collapsed, and some fluid appeared in the Douglas pouch.

SECONDARY OUTCOMES:
Serum progesterone | Day 8 post hCG injection
  Serum progesterone will be measured on day 8 post hCG injection, ovulation will be confirmed if the serum progesterone level is ≥ 5 ng/ml.
Clinical pregnancy | 14 days after hCG administration
  Pregnancy test will be done in the form of testing the level of beta hCG in the blood after 14 days once the success of the ovulation process has been confirmed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics and gynaecology, faculty of medicine, Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
L-Carnitine and Clomiphene Citrate for induction of ovulation in women with Polycystic Ovary Syndrome